CLINICAL TRIAL: NCT03045133
Title: QUALITY OF RECOVERY AFTER INTRAOPERATIVE MORPHINE OR METHADONE IN PATIENTS UNDERGOING LAPAROSCOPIC CHOLECYSTECTOMY
Brief Title: QUALITY OF RECOVERY AFTER INTRAOPERATIVE MORPHINE OR METHADONE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidade Catolica de Sao Paulo (Other)
Responsible Party: Principal Investigator, Eduardo Toshiyuki Moro, Professor, Pontificia Universidade Catolica de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PUCSP 050539/2016
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Pain, Postoperative; Nausea and Vomiting, Postoperative
Keywords: Postoperative pain; Postoperative nausea and vomiting; Quality of recovery; QoR-40; Total intravenous anesthesia
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Methadone; Morphine

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blinded trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Group assignments were sealed in sequentially numbered opaque envelopes that were opened after patient inclusion in the study. All care providers, researchers, and patients were blinded to group assignments. Study 10-mL syringes will be prepared by an anesthesiologist independent of the study. Methadone 0.1 mg.kg-1 (made up to 10 mL with normal saline) or morphine 0.1 mg.kg-1 (made up to 10 mL with normal saline) will be drawn into each syringe which will be offered to the anesthesia provider after the opaque envelope is opened.
  The baseline QoR-40 questionnaire will be provided to subjects after informed consent is obtained in the preoperative holding area and 24 hours after surgery by a blinded investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MT group (Active Comparator): Immediately after the induction of anesthesia, patients will receive intravenously methadone 0.1 mg/kg
  Interventions: Drug: Methadone
- MF group (Active Comparator): Immediately after the induction of anesthesia, patients will receive intravenously morphine 0.1 mg/kg
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Methadone — Immediately after the induction of anesthesia, patients will receive intravenously methadone 0.1 mg/kg
  Arms: MT group
Drug: Morphine — Immediately after the induction of anesthesia, patients will receive intravenously morphine 0.1 mg/kg
  Arms: MF group

SUMMARY:
Introduction. Despite the advantages associated with the use of remifentanil during total intravenous anesthesia (TIVA), it has been observed a frequent difficulty in the control of postoperative pain due to the risk of developing hyperalgesia and acute tolerance associated with the administration of this opioid. There is evidence that NMDA receptors are involved in the development of these changes. Methadone is an opioid that exhibits analgesic potency similar to that of morphine but has NMDA antagonist activity and longer duration of action as additional features. The objective of the study was to evaluate the quality of recovery (QoR40) of patients undergoing TIVA for laparoscopic cholecystectomy and who received morphine or methadone to control postoperative pain. Methods. Patients aged 18 to 65 years, physical status ASA I and II, submitted to total venous anesthesia (propofol and remifentanil) for laparoscopic cholecystectomy and eligible to participate in this prospective and randomized clinical study will be evaluated. After induction of anesthesia, patients will receive a solution containing 0.1 mg.kg-1 morphine (MF group) or 0.1 mg.kg-1 methadone (MT group). Data on the presence of pain, nausea, vomiting, tremor, drowsiness, presence of SpO2 <92%, even with O2 face mask (5 L.min-1) and length of stay will be recorded at PACU. The pain will be evaluated every 15 minutes on a verbal numerical scale (ENV) from 0 to 10. E.v. morphine 0.1 mg.kg-1 (MF group) or methadone 0.1 mg.kg-1 (MT group) will be administered every 15 minutes to obtain the score below 3. After discharge from the PACU, all patients will receive intravenous ketoprofen every 12 hours and dipyrone every 6 hours. For cases where the patient considers the analgesic regimen insufficient, tramadol (100 mg) will be administered intravenously at 8-hour intervals. The consumption of analgesics, the intensity of pain, the occurrence of nausea, vomiting and other complications in the ward will be recorded. The application of the questionnaire (QoR40) will be performed in the ward the morning after the surgery by a medical student.

DETAILED DESCRIPTION:
We hypothesized that methadone treatment would beneficially affect patient-perceived quality of recovery after laparoscopic cholecystectomy under total intravenous anesthesia. The primary outcome was assessed using the Quality of Recovery Questionnaire (QoR-40), a 40-item quality of recovery scoring system, on postoperative day (POD) 1. In addition, the effects of both opioids on early clinical recovery variables, such as the time to eye opening, the occurrence of nausea and vomiting, pain score, use of analgesics, and length of PACU stay, were determined.

Methods. This randomised trial was approved by the Research Ethics Committee of the School of Medical and Health Sciences, Pontifical Catholic University of São Paulo.

Study sequence No premedication will be applied to the patients. Patients´ preoperative data including age, gender, physical status and, BMI will be collected. Subjects will be randomized using a computer-generated (www.random.org) table of random numbers into 2 groups: MT (methadone 0.1 mg.kg-1) or MF (morphine 0.1 mg.kg-1). Group assignments were sealed in sequentially numbered opaque envelopes that were opened after patient inclusion in the study. All care providers, researchers, and patients were blinded to group assignments. Two study 10-mL syringes will be prepared by an anesthesiologist independent of the study. Syringe 1 to be used during intraoperative phase and syringe 2 as a rescue for postoperative pain. Methadone 0.1 mg.kg-1 (made up to 10 mL with normal saline) or morphine 0.1 mg.kg-1 (made up to 10 mL with normal saline) will be drawn into each syringe which will be offered to the anesthesia provider after the opaque envelope is opened.

Anesthetic and Surgical Management After arrival in the operating room, standard ASA monitors will be applied. Lidocaine (30 mg) will be administered intravenously immediately after venoclysis. After anesthesia induction, capnographic monitoring will be added. Anesthesia will be induced with remifentanil 0.5 µg.kg-1.min-1 over three minutes followed by propofol 2.0 mg. kg-1. Rocuronium 0.6 mg.kg-1 will be administered to facilitate tracheal intubation. Anesthetic maintenance will be achieved with a continuous infusion of remifentanil 0.3 µg.kg-1.min-1 and propofol 4 to 6 mg. kg-1. h-1. Ventilation will be controlled mechanically to maintain an end-tidal carbon dioxide concentration of 30-40 mmHg using a 50% oxygen-air gas mixture. Immediately after the induction of anesthesia, patients will receive intravenously: MT group - Methadone 0.1 mg/kg or MF group - morphine 0.1 mg/kg. Patients who exhibit reductions in systolic arterial pressure (SAP) greater than 30% or heart rate (HR) reductions to less than 50 bpm will be given ephedrine (10 mg) and atropine (0.5 mg), respectively. Normal saline will be used for fluid replacement therapy at a rate of 500 ml throughout the first 30 minutes, and, then, 2 ml/kg/h until the end of the surgical procedure. All of the participants will receive dexamethasone (8 mg) and ketoprofen (100 mg) at the onset of surgery and ondansetron (4 mg) and dipyrone (1 g). Residual neuromuscular blockade will be antagonized by atropine (0.01 mg/ kg) and neostigmine (0.015 mg/kg). Extubation will be performed after awakening. The time elapsed from discontinuation of the anesthetics until the eye opening will be registered.

When stable vital signs and respiration are confirmed, all patients will be transferred to the post-anesthesia care unit (PACU). Early recovery times includes time to eye opening (time from the discontinuation of anaesthetics to eye opening) and time to Aldrete score ≥ 9. Data related to the occurrence of pain, nausea and vomiting at the PACU will be recorded. Pain will be assessed while at rest and after asking the subjects to cough, every 15 minutes using a 0-10 numeric pain rating scale (NRS), where zero meant no pain and 10 the worst imaginable pain. When stable vital signs and respiration are confirmed, all patients will be transferred to the post-anesthesia care unit (PACU). Early recovery times includes time to eye opening (time from the discontinuation of anaesthetics to eye opening) and time to Aldrete score ≥ 9. Data related to the occurrence of pain, nausea and vomiting at the PACU will be recorded. Pain will be assessed while at rest and after asking the subjects to cough, every 15 minutes using a 0-10 numeric pain rating scale (NRS), where zero meant no pain and 10 the worst imaginable pain. One or two mL from the solution previously prepared (Syringe 2) will be administered intravenously every 15 minutes to maintain the pain score below 3 (1 mg when the pain score is <7 and 2 mg when it is ≥7). Following discharge from the PACU (minimum stay 60 minutes and Aldrete score ≥ 9), all of the participants will receive ketoprofen (100 mg) every 12 hours and dipyrone (30 mg.kg-1, maximum 1 g) every six hours intravenously. Whenever patients judge that their analgesia is insufficient, tramadol (100 mg) will be administered intravenously at eight-hour minimum intervals. Postoperative nausea and vomiting (PONV) will be treated with ondansetron (4 mg) intravenously. An investigator who will be blinded to group assignment will collect all postoperative outcome data 24 hours after surgical procedure. Subjects will rate the higher score of pain (NRS) during the hospital ward stay. Tramadol consumption and the number of nausea and vomiting episodes will also be recorded. These findings will be confirmed with the ward nursing staff. All subjects will stay at hospital for at least 24 hours.

Data Collection The baseline QoR-40 questionnaire will be provided to subjects after informed consent is obtained in the preoperative holding area and 24 hours after surgery by a blinded investigator. The QoR-40 questionnaire assesses five dimensions of recovery (physical comfort - 12 items; emotional state - 7 items; physical independence - 5 items; physiological support - 7 items; and pain - 7 items). Each item is rated on a five-point Likert scale: none of the time, some of the time, usually, most of the time, and all the time. The total score on the QoR-40 ranges from 40 (poorest quality of recovery) to 200 (best quality of recovery). The primary outcome of interest will be the QoR-40 score, however the following data will also be recorded: age, gender, physical status, BMI, and length of PACU stay.

Statistical Analysis The sample size was calculated considering 90% power to detect a 10-point difference in QoR-40, which indicated the need to include 31 participants in each group. Taking possible losses into consideration, the final sample included 70 patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II, who will be scheduled to undergo laparoscopic cholecystectomy at Santa Lucinda Hospital

Exclusion Criteria:

* Patients who (i) refuse to participate in the study; (ii) are not able to communicate due to alterations in the level of consciousness, or neurologic, or psychiatric disease; - present with contraindication to any of the drugs used in the present study
* have history of alcohol or drug abuse
* present a body mass index (BMI) ≥ 40 will be excluded.
* Reasons for exclusion after randomization will be protocol violations or if the surgical procedure changes from a laparoscopic to an open approach.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2016-07-20 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Quality of recovery (QoR-40) | 24 hours
  The baseline QoR-40 questionnaire will be provided to subjects after informed consent is obtained in the preoperative holding area and 24 hours after surgery by a blinded investigator. The QoR-40 questionnaire assesses five dimensions of recovery (physical comfort - 12 items; emotional state - 7 items; physical independence - 5 items; physiological support - 7 items; and pain - 7 items). Each item is rated on a five-point Likert scale: none of the time, some of the time, usually, most of the time, and all the time. The total score on the QoR-40 ranges from 40 (poorest quality of recovery) to 200 (best quality of recovery).

SECONDARY OUTCOMES:
Time to eye opening | 30 minutes
  The time elapsed from discontinuation of the anesthetics until the eye opening
Postoperative pain (PACU) | 2 hours
  Pain will be assessed while at rest and after asking the subjects to cough, every 15 minutes using a 0-10 numeric pain rating scale (NRS), where zero meant no pain and 10 the worst imaginable pain.
Postoperative pain (Ward) | 24 hours
  Subjects will rate the higher score of pain (NRS) during the hospital ward stay
Tramadol consumption | 24 hours
  Consumption, or not, of tramadol during the hospital ward stay
Postoperative nausea and vomiting | 24 hours
  Number of episodes of vomiting or the occurrence of nausea
Time of PACU staying | 3 hours
  Time required to meet and achieve PACU discharge criteria (Aldrete 9)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo T Moro, Professor, Principal Investigator — PUC São Paulo University
Locations (1):
- Santa Lucinda Hospital, Sorocaba, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No